CLINICAL TRIAL: NCT03610438
Title: A Phase IIA Study of Feasibility and Effectiveness of Inotuzumab Ozogamicin (IO) in Adult Patients With B-Cell Acute Lymphoblastic Leukemia With Positive Minimal Residual Disease Before Any Hematopoietic Stem Cell Transplantation
Brief Title: Feasibility and Effectiveness of Inotuzumab Ozogamicin in B-Cell Acute Lymphoblastic Leukemia
Acronym: ALL2418
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALL2418; 2018-003006-32 (EudraCT Number)
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Acute Lymphoid Leukemia
Keywords: Acute Lymphoid Leukemia; Inotuzumab Ozogamicin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Intervention Model Description: The study is divided in two cohorts; cohort 1 will enroll 38 Ph+ patients, cohort 2 will enroll 38 Ph- patients, as defined with statistical analysis. The two cohorts will have the same treatment, with the exception of short term and long term maintenance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will entroll 38 Ph+ patients
  Interventions: Drug: Inotuzumab Ozogamicin (IO)
- Cohort 2 (Experimental): Cohort 2 will enroll 38 Ph- patients
  Interventions: Drug: Inotuzumab Ozogamicin (IO)

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin (IO) — After course 1 MRD will be evaluated:
  - patients MRD negative will enter into short maintenance or long maintenance according to investigator choice. After 4 to 12 weeks in short maintenance patient will undergo SCT, otherwise, patients will enter long maintenance.
  Arms: Cohort 1
Drug: Inotuzumab Ozogamicin (IO) — After course 2 MRD will be evaluated; patients MRD negative will enter into short maintenance or long maintenance by investigator choice. After 4 to 12 weeks in short maintenance patient will undergo SCT, otherwise, patients will enter long maintenance.
  Arms: Cohort 2

SUMMARY:
This is a multi-center, phase 2A exploratory study of feasibility and effectiveness of Inotuzumab Ozagomicin in adult patients with Acute Lymphoid Leukemia (ALL) with positive minimal residual disease before any hematopoietic stem cell transplantation.

The study is divided in two cohorts; cohort 1 will enroll 38 Ph+ patients, cohort 2 will enroll 38 Ph- patients, as defined with statistical analysis. The two cohorts will have the same treatment, with the exception of short term and long term maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Ph+ ALL with p190 or p210 detectable and measurable (at least 10-4 x10000 ABL) after at least 3 months of any therapy, or the failure of at least 2 TKI.
* Ph- ALL with detectable and measurable IG specific transcript after at least 2 courses of previous therapy.
* Age ≥ 18 years old.
* ECOG ≤ 2.

Exclusion Criteria:

* More than 5% of BM blasts.
* WHO performance status ≤ 50% (Karnofsky) or ≥ 3 (ECOG).
* Active HBV or HCV hepatitis, or AST/ALT ≥ 2.5 x ULN and bilirubine ≥ 1.5 x ULN.
* Evidence of liver fibrosis, portal hypertension or other clinically relevant liver abnormalities at screening liver ultrasonography.
* History of alcohol abuse.
* Burkitt lymphoma and active CNS leukemia. Patients with previuos neurological toxicitiy as well co-morbidity will be carefully evaluated for enrolment.
* Ongoing or active infections.
* Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL). Clinically significant, uncontrolled, or active cardiovascular disease.
* Uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
* Creatinine level > 2.5mg/dl or Glomerular Filtration Rate (GFR) < 20 ml/min or proteinuria > 3.5 g/day.
* Documented inherited protrombotic disorders
* Patients who have received any investigational drug ≤ 4 weeks.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention or with a life expectancy due to other malignancy <6 months.
* Patients that have received Inotuzumab or Anti CD22 directed therapies before
* Patients with known hereditary coagulopathy
* Patient that received during their life diagnosis of VOD or had ongoing VOD
* Patients who are pregnant or breastfeeding and adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of induction therapy). Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 4 months following discontinuation of study drugs.
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients obtaining a negative Minimal Residual Disease (MRD) | Two years after study entry.

SECONDARY OUTCOMES:
Number of patients alive | Two years from start of treatment.
Number of adverse events in MRD positive patients | Two years after study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Study Chair — Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST Italy; Fabio Ciceri, Study Director — Istituto S. Raffaele, Milan, Italy Giuseppe Saglio, Institute of Hematology, Ospedale Mauriziano, Turin, Italy
Locations (30):
- Italy (30):
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona- Sod Clinica Ematologica, Ancona
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - As Dell'Alto Adige, Ospedale Centrale Di Bolzano - Ematologia E Centro Trapianto Midollo Osseo, Bolzano
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Aso S. Croce E Carle - Cuneo - Sc Ematologia, Cuneo
  - Irccs Aou San Martino - Genova - Uo Clinica Ematologica, Genova
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - I.R.S.T. Srl Irccs - Meldola - Sc Oncologia Medica, Meldola
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Istituto Europeo Di Oncologia Irccs - Milano - Divisione Di Oncoematologia, Milan
  - Ao Di Rilievo Nazionale Antonio Cardarelli - Napoli - Uoc Ematologia Con Trapianto Di Midollo, Napoli
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli" Po E. Morelli - Reggio Calabria - Uoc Ematologia, Reggio Calabria
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Unità Operativa Di Ematologia - Presidio Ospedaliero Di Treviso - Azienda Ulss N.2 Marca Trevigiana, Treviso
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it